CLINICAL TRIAL: NCT05355207
Title: Phase 1 Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of TRL1068 in Subjects With Acute Exacerbation of Chronic Rhinosinusitis
Brief Title: Study to Evaluate Safety and Activity of TRL1068 in Chronic Rhinosinusitis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Trellis Bioscience LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRL1068-104
Record Dates: First submitted 2022-04-18; First posted 2022-05-02 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps
Keywords: biofilm; antibiotic-resistant infections
MeSH Terms: interventions — TRL1068

STUDY DESIGN:
Intervention Model Description: single group, all subjects will receive 15 mg/kg of TRL1068 on Day 1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TRL1068 (Experimental): all subjects will receive a single intravenous dose of 15 mg/kg of TRL1068 on Day 1
  Interventions: Drug: TRL1068

INTERVENTIONS:
Drug: TRL1068 — A human IgG1κ (G1m1,17 (z,a); Km3 allotype) monoclonal antibody

SUMMARY:
TRL1068 is expected to eliminate the pathogen-protecting biofilm in Chronic Rhinosinusitis, thus making these bacteria substantially more susceptible to established antibiotic treatment regimens. This initial study is to assess overall safety and pharmacokinetics (PK) of TRL1068. The goal of the development program is to demonstrate effectiveness of TRL1068 in difficult to treat bacterial infections such as in CRS.

DETAILED DESCRIPTION:
Chronic rhinosinusitis with nasal polyps (CRSwNP) is associated with significant morbidity and decreased quality of life. Defects in the epithelial cell barrier, increased exposure to pathogenic and colonized bacteria, and dysregulation of the host immune system are all thought to play prominent roles in disease pathogenesis. Colonization with S. aureus or P. aureus are associated with recalcitrant disease and biofilm formation, making eradication difficult.

Distribution of topical solutions in the unoperated sinuses has been observed to be less than 2% of the total irrigation volume, with almost no penetration in the frontal and sphenoid sinuses. For those patients with mucosal edema from infection and chronic inflammation, distribution is probably significantly less when applied topically. Intravenously administered TRL1068 is expected to achieve effective anti-biofilm levels throughout the sinonasal space for several weeks. TRL1068 is a monoclonal human antibody that rapidly eliminates biofilm at very low concentrations, thus making the targeted bacterial pathogens substantially more sensitive to standard of care antibiotic treatment regimen and greatly accelerating clinical improvement and potential for bacterial eradication.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 85 years, inclusive
2. Diagnosis of chronic rhinosinusitis with:

   1. Acute exacerbation of CRSwNP with increased sinonasal discharge OR
   2. Acute exacerbation post-functional endoscopic sinus surgery (FESS) with increased sinonasal discharge AND
   3. Sinonasal culture positive for SA or PA without concomitant fungal infection in culture or PCR
3. Symptoms and culture results justify initiation of topical and/or systemic antibiotic treatment
4. Willing and able to provide written informed consent
5. Willing to perform and comply with all study procedures including attending clinic visits as scheduled
6. Men and women of child bearing potential (WOCBP) must be willing to practice a highly effective method of contraception that may include, but is not limited to, abstinence, sex only with persons of the same sex, monogamous relationship with vasectomized partner, vasectomy, hysterectomy, bilateral tubal ligation, licensed hormonal methods, intrauterine device (IUD), or use of spermicide combined with a barrier method (e.g., condom, diaphragm) for 28 days before receiving the investigational product (IP) and through Day 50.

Exclusion Criteria:

1. Active malignancy, or history of malignancy or chemotherapy within the past 2 years other than history of localized or surgical removal of focal skin cancer, or cervical cancer in situ treated successfully in the past by local treatment (including but not limited to cryotherapy or laser therapy) or by hysterectomy
2. Any chronic or acute bacterial infection other than acute exacerbation of CRS
3. Concomitant intrasinal culture or 16S PCR indicative of concomitant fungal infection
4. Allergic fungal rhinosinusitis, characterized by elevated antifungal IgE and eosinophilic mucus
5. Receiving or recently received another investigational drug (within 30 days of Day 1, or 5 half-lives of the investigational drug, whichever is longer)
6. Received a COVID-19 vaccine or booster within 14 days of planned Day 1 or planned COVID-19 vaccination within 14 days after Day 1
7. Positive serum test for pregnancy, pregnant, or nursing women
8. History of drug or alcohol abuse that, in the opinion of the Investigator, would interfere with the subject's ability to comply with the study requirements
9. Any other comorbidity or condition that, in the opinion of the Investigator would make the subject unsuitable for the study or unable to comply with the study requirements

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of abnormal physical exam findings | 6 weeks
  Clinically-significant abnormal physical exam findings will be reviewed
Incidence of abnormal serum chemistries and hematology | 6 weeks
  Clinically-significant abnormal laboratory results will be reviewed
Incidence of abnormal vital signs (temperature) | 6 weeks
  Clinically-significant abnormal temperatures will be reviewed
Incidence of abnormal vital signs (blood pressure) | 6 weeks
  Clinically-significant abnormal blood pressures will be reviewed
Incidence of abnormal vital signs (heart rate) | 6 weeks
  Clinically-significant abnormal heart rates will be reviewed
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 7 weeks
  reported AEs and SAEs will be reviewed
Characterize the pharmacokinetics (PK) of TRL1068 in serum (Cmax) | 6 weeks
  Individual subject TRL1068 Cmax in serum will be determined by ELISA and derived PK parameters will be summarized using descriptive statistics.
Characterize the pharmacokinetics (PK) of TRL1068 in serum (Cmin) | 6 weeks
  Individual subject TRL1068 Cmin in serum will be determined by ELISA and derived PK parameters will be summarized using descriptive statistics.
Characterize the pharmacokinetics (PK) of TRL1068 in serum (Tmax) | 6 weeks
  Individual subject TRL1068 Tmax in serum will be determined by ELISA and derived PK parameters will be summarized using descriptive statistics.
Characterize the pharmacokinetics (PK) of TRL1068 in serum (AUCLAST) | 6 weeks
  Individual subject TRL1068 AUCLAST in serum will be determined by ELISA and derived PK parameters will be summarized using descriptive statistics.
Characterize the pharmacokinetics (PK) of TRL1068 in serum (AUCINF) | 6 weeks
  Individual subject TRL1068 AUCINF in serum will be determined by ELISA and derived PK parameters will be summarized using descriptive statistics.
Characterize the pharmacokinetics (PK) of TRL1068 in intrasinal concentrations (Cmax) | 6 weeks
  Individual subject TRL1068 Cmax intrasinal will be determined by ELISA and derived PK parameters will be summarized using descriptive statistics.
Characterize the pharmacokinetics (PK) of TRL1068 in intrasinal concentrations (Cmin) | 6 weeks
  Individual subject TRL1068 Cmin intrasinal will be determined by ELISA and derived PK parameters will be summarized using descriptive statistics.
Characterize the pharmacokinetics (PK) of TRL1068 in intrasinal concentrations (Tmax) | 6 weeks
  Individual subject TRL1068 Tmax intrasinal will be determined by ELISA and derived PK parameters will be summarized using descriptive statistics.
Characterize the pharmacokinetics (PK) of TRL1068 in intrasinal concentrations (AUCLAST) | 6 weeks
  Individual subject TRL1068 AUCLAST intrasinal will be determined by ELISA and derived PK parameters will be summarized using descriptive statistics.
Characterize the pharmacokinetics (PK) of TRL1068 in intrasinal concentrations (AUCINF) | 6 weeks
  Individual subject TRL1068 AUCINF intrasinal will be determined by ELISA and derived PK parameters will be summarized using descriptive statistics.
Characterize the pharmacodynamics (PD) of TRL1068 (time to resolution of bacterial pathogen infection) | 6 weeks
  Cultures will be tested for bacterial pathogen presence by bacterial culture and/or PCR assessment. Time to resolution of bacterial pathogen infection is defined as the number of days from start of current acute exacerbation to the day when testing by bacterial culture and/or PCR assessment are reported as negative. Descriptive statistics will be performed including mean, median and confidence interval.
Characterize the pharmacodynamics (PD) of TRL1068 (time to resolution of signs and symptoms of acute exacerbation) | 6 weeks
  Patients will be evaluated for signs and symptoms of acute exacerbation using SNOT-22 scoring. Time to resolution of signs and symptoms of acute exacerbation is defined as the day when the SNOT-22 score is back to pre-acute exacerbation score.
Assess the immunogenicity of TRL1068 as measured by anti-drug antibodies (ADAs) | 6 weeks
  Anti-drug antibodies (ADA), i.e. anti-TRL1068 antibodies in serum will determined by electrochemiluminescence assay

SECONDARY OUTCOMES:
Assess the incidence of improvement of baseline symptoms of chronic rhinosinusitis (CRS) after intravenous TRL1068 | 7 weeks
  signs and symptoms will be measured using the SNOT-22
Assess time to improvement of baseline symptoms of CRS as compared with previous duration of acute exacerbations | 7 weeks
  signs and symptoms will be measured using the SNOT-22 and compared with historical data

OTHER OUTCOMES:
Assess the effects of treatment on the intrasinal microbiome | 6 weeks
  intrasinal culture and PCR results will be reviewed

IPD SHARING:
Plan to Share IPD: Yes
We plan to make the Clinical Protocol and SAP available on Protocols.io (https://www.protocols.io/) before trial recruitment is complete.
Supporting Information: Study Protocol, SAP
Time Frame: Before trial recruitment is complete on Protocols.io (https://www.protocols.io/)
Access Criteria: available

REFERENCES:
- [Background] Estelles A, Woischnig AK, Liu K, Stephenson R, Lomongsod E, Nguyen D, Zhang J, Heidecker M, Yang Y, Simon RJ, Tenorio E, Ellsworth S, Leighton A, Ryser S, Gremmelmaier NK, Kauvar LM. A High-Affinity Native Human Antibody Disrupts Biofilm from Staphylococcus aureus Bacteria and Potentiates Antibiotic Efficacy in a Mouse Implant Infection Model. Antimicrob Agents Chemother. 2016 Mar 25;60(4):2292-301. doi: 10.1128/AAC.02588-15. Print 2016 Apr. PMID 26833157
- [Background] Xiong YQ, Estelles A, Li L, Abdelhady W, Gonzales R, Bayer AS, Tenorio E, Leighton A, Ryser S, Kauvar LM. A Human Biofilm-Disrupting Monoclonal Antibody Potentiates Antibiotic Efficacy in Rodent Models of both Staphylococcus aureus and Acinetobacter baumannii Infections. Antimicrob Agents Chemother. 2017 Sep 22;61(10):e00904-17. doi: 10.1128/AAC.00904-17. Print 2017 Oct. PMID 28717038